CLINICAL TRIAL: NCT05188391
Title: A Novel Examination Method for Deltoid Injuries: Deltoid Gap Sign
Brief Title: A New Method for Deltoid Ruptures: Gap Sign
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Goztepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Esat UYGUR, Assoc.Prof.M.D., Goztepe Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2021-04
Record Dates: First submitted 2021-11-30; First posted 2022-01-12 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Ankle Fractures; Ligament Rupture; Ligament Injury
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Physicians who will perform the examination will not know other physicians' decisions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Positive Group (Rupture and Gap Sign are both positive) (Other): Rupture and Gap Sign are both positive
  Interventions: Diagnostic Test: Deltoid Gap Sign
- Rupture Positive Group (Rupture positive but Gap Sign is negative) (Other): Rupture positive but Gap Sign is negative
  Interventions: Diagnostic Test: Deltoid Gap Sign
- Gap Sign Positive Group (No rupture exists but Gap Sign is positive) (Other): No rupture exists but Gap Sign is positive
  Interventions: Diagnostic Test: Deltoid Gap Sign
- Negative Group (Rupture and Gap sign are both negative) (Other): Rupture and Gap sign are both negative
  Interventions: Diagnostic Test: Deltoid Gap Sign

INTERVENTIONS:
Diagnostic Test: Deltoid Gap Sign — At first deltoid sign test will be performed and the result of the test will be noted for the patients who are already scheduled open medial ankle surgery due to diagnosed as ankle fracture. During the open surgery, the test results will be evaluated.
  Other Names: Open (visual) Examination of the ligament

SUMMARY:
"Deltoid Gap Sign" which would be a new method of examination for deltoid ligament injuries will be investigated. It will be analyzed if it is correlated with the external rotation stress test. The study is designed as a blinded, comparative and prospective trial.

DETAILED DESCRIPTION:
Ankle fracture patients who applied to our clinic agreed to be included in the study and underwent surgical intervention will participate in the study. The pediatric age group will not be included in the study, since deltoid ligament tears are not common in ankle fractures in pediatric age. However, since this fracture can also be seen in pregnant women, if there is a pregnant patient who will require surgical treatment, they can be included in the study.

"Deltoid Gap Sign" which is the main subject of this study, will be performed in patients firstly at patients' ward i) without pre-operative anesthesia, secondly at operating theatre ii) under anesthesia before the operation. The examination will be carried out by two different physicians and the opinion of both physicians will be noted. Physicians will be blinded and will not know others' decisions.

External rotation stress test (ERST) in dorsiflexion, which is another examination method accepted in the literature in the evaluation of the deltoid ligament, will also be performed by two physicians and the opinions of the physicians will be noted. ERST will be analyzed under fluoroscopy control.

After the examination, open surgery will be performed around the medial malleolus. It will be noted whether the deltoid ligament was injured (ruptured/ not ruptured), which fibers of the deltoid ligament (superficial/deep/superficial + deep fibers) were ruptured.

Statistical ratios such as positive predictive value, negative predictive value, sensitivity, specificity, and likelihood ratio will be calculated based on the results obtained.

Deltoid gap sign will be checked whether it is correlated with ERST and the results will be compared with the ERST.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had operated on because of ankle trauma
* Patients who had been performed an open surgery at the medial malleolus region
* Patients with Maisonneuve fractures

Exclusion Criteria:

* Medial malleolus fractures
* Talus fractures
* Patients in pediatric age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2023-08-04 (Estimated); Study Completion 2023-12-04 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the Gap Sign | 24 hours
  Gap Sign will be recorded either positive or negative after performing Deltoid Gap Sign. During the open surgery, the rupture of the ligament will be evaluated again. Then sensitivity of Gap Sign will be calculated using Chi Square test.

SECONDARY OUTCOMES:
Specificity of the Gap Sign | 24 hours
  Gap Sign will be recorded either positive or negative after performing Deltoid Gap Sign. During the open surgery, the rupture of the ligament will be evaluated again. Then specificity of Gap Sign will be calculated using Chi Square test.
Likelihood ratios of the Gap Sign | 24 hours
  Gap Sign will be recorded either positive or negative after performing Deltoid Gap Sign. During the open surgery, the rupture of the ligament will be evaluated again. Then likelihod ratios of Gap Sign will be calculated using Chi Square test.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medeniyet University.Göztepe State Hospital, Istanbul, Kadıkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No